CLINICAL TRIAL: NCT06259500
Title: Generation and Analysis of Patient-derived Stem Cell Models of Hypothalamic Neurons and Microglia in Anorexia Nervosa
Brief Title: Patient-derived Stem Cell Models of Anorexia Nervosa
Acronym: ANSTEM
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ida AK Nilsson, Associate Professor, Karolinska Institutet
Other Study IDs: 2019 00170
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-03

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- anorexia nervosa
  Interventions: Other: observational
- healthy controls
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — Profiling the function of iPSC derived Arcuate neurons and PBMC derived microglia

SUMMARY:
Experimental and genetic data, as well as brain imaging, support a role of the hypothalamic Arcuate nucleus neurons and their communication with surrounding microglia in anorectic conditions, but it has until recently not been possible to explore these cells at a molecular level in anorexia nervosa (AN) patients. This attributed to the obvious lack of valid tissue and non-invasive imaging techniques of high enough resolution. Stem cell models have evolved as a useful tool for the exploration of other neuropsychiatric disorders with a comparably high genetic contribution as AN. The investigators will here use patient-derived induced pluripotent stem cells (iPSCs) to profile Arc neurons and peripheral blood mononuclear cell (PBMC) derived microglia in AN, thus defining molecules to explore as drug targets.

ELIGIBILITY:
Inclusion Criteria anorexia nervosa:

* female
* 18-45 years of age
* AN restrictive diagnosis as main diagnosis
* more than 5 years duration

Exclusion Criteria anorexia nervosa:

-

Inclusion Criteria healthy control:

* female
* 18-45 years of age
* BMI 18,5 - 25

Exclusion Criteria healthy control:

* own or family member with eating disorder diagnosis
* own or family member with autism diagnosis

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only female participants
Study Population: Patients recruited from specialised care unit Controls from community
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Microglia function and transcriptomic profiling | 2025
  phagocytic and immune activation capacity and whole transcriptomic profiling, anorexia nervosa vs healthy controls
Arcuate neuron function and transcriptomic profiling | 2026
  Electrical activity, transmitter release and whole transcriptomic profiling of iPSC derived Arcuate neurons, anorexia nervosa vs healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No